CLINICAL TRIAL: NCT01527760
Title: Effectiveness of Viscum Album Mother Tincture as an Anti-hypertensive in Essential Hypertension. One Group Pretest Posttest Design
Brief Title: Effectiveness of Viscum Album Mother Tincture as an Anti-hypertensive in Essential Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fr Muller Homoeopathic Medical College (Other)
Collaborators: Rajiv Gandhi University of Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Kurian P J, Lecturer, Fr Muller Homoeopathic Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGUHS2010
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Hypertension
Keywords: Essential Hypertension; Viscum album mother tincture; one group pretest post-test study
MeSH Terms: conditions — Hypertension; Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Viscum album ethanolic extract manufactured according to Homoeopathic pharmacopoeia of India (H.P.I.) — Ten drops of Drug in 30 ml of distilled water with a frequency of three times a day for a duration of 12 weeks

SUMMARY:
To estimate the effectiveness of Viscum album Homoeopathic mother tincture in Essential Hypertension by conducting clinical trial in moderate hypertensive patients for a period of six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension at the range 180-120 mm of Hg for Systole &
* 110-80 mm of Hg for Diastole

Exclusion Criteria:

* Patients who are on ACEI / ARB for Hypertension
* Diseases in which life expectancy is less than six months
* Secondary hypertension
* CHD
* Family History of Mental Illness like Anxiety or depression.
* Nasal Congestion

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in Systolic and Diastolic blood pressure. | 12 weeks

SECONDARY OUTCOMES:
Change in Serum Cholesterol | 12 weeks
Change in Serum Triglycerides | 12 weeks
Change in Serum LDH | 12 weeks
Change in Serum Urea | 12 weeks
change in Serum CKMB | 12 weeks and 16 weeks
  The blood sample was collected at the end of 12 weeks of medication followed by a drug free period of 4 weeks.The blood sample was collected again at the end of 4 weeks of drug free period to ascertain serum CKMB.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kurian P John, MD, Principal Investigator — Fr Muller Homoeopathic Medical College
Locations (1):
- Fr Muller Homoeopathic Medical College Hospital, Mangalore, Karnataka, India

REFERENCES:
- [Derived] Poruthukaren KJ, Palatty PL, Baliga MS, Suresh S. Clinical evaluation of Viscum album mother tincture as an antihypertensive: a pilot study. J Evid Based Complementary Altern Med. 2014 Jan;19(1):31-5. doi: 10.1177/2156587213507726. Epub 2013 Nov 5. PMID 24647376